CLINICAL TRIAL: NCT02773758
Title: Short Term Clinical Study Investigating the Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity
Brief Title: Study to Investigate the Efficacy of an Occluding Dentifrice in Providing Relief From Dentine Hypersensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205201
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stannous Fluoride Dentifrice (Experimental): Participants will be instructed to topically dose a dry toothbrush with a full strip of toothpaste, then brush each of the two selected sensitive test teeth first, followed by the whole mouth thoroughly for at least 1 minute twice daily (morning and evening). Participants will be permitted to rinse with tap water.
  Interventions: Other: Stannous Fluoride Dentifrice
- Sodium monofluorophosphate Dentifrice (Other): Participants will be instructed to topically apply a full brush head of toothpaste to a dry toothbrush, then brush the whole mouth thoroughly for at least 1 minute. Participants will be permitted to rinse with tap water.
  Interventions: Other: Sodium monofluorophosphate Dentifrice

INTERVENTIONS:
Other: Stannous Fluoride Dentifrice — Experimental dentifrice containing 0.454%w/w stannous fluoride (1100ppm fluoride)
  Arms: Stannous Fluoride Dentifrice
Other: Sodium monofluorophosphate Dentifrice — Dentifrice containing 0.76% w/w sodium monofluorophosphate (1000ppm fluoride)
  Arms: Sodium monofluorophosphate Dentifrice

SUMMARY:
This will be a single centre, two week, randomised, examiner blind, two treatment arm, parallel design, stratified (by maximum baseline Schiff sensitivity score of the two selected test teeth), controlled study, in participant with at least two sensitive teeth that meet the study criteria at the Screening and Baseline visits. The study will be conducted in participants in good general health, with pre-existing self-reported and clinically diagnosed tooth sensitivity at screening.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged 18-65 years inclusive.
* Good general and mental health with:

No clinically significant and relevant abnormalities of medical history or oral examination.

Absence of any condition that would impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.

* Self-reported history of dentinal hypersensitivity (DH) lasting more than six months but not more than 10 years.
* Minimum of 20 natural teeth.
* Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria at screening: Signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR).

Tooth with MGI score =0 adjacent to the test area (exposed dentine) only and a clinical mobility of ≤1.

Tooth with signs of sensitivity measured by qualifying evaporative air assessment (yes[Y]/No[N] response).

* Minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars), that meet all of the following criteria at screening:

Tooth with signs of sensitivity, measured by response to a qualifying tactile stimulus (Yeaple ≤ 20g) and evaporative air assessment (Schiff sensitivity score ≥ 2).

Exclusion Criteria:

* Women who are breast-feeding, known to be pregnant or who are intending to become pregnant over the duration of the study.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Previous participation in this study or participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Recent history (within the last year) of alcohol or other substance abuse.
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes or causing xerostomia.
* Dental prophylaxis within 4 weeks of Screening.
* Tongue or lip piercing or presence of dental implants.
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening.
* Teeth bleaching within 8 weeks of Screening.
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening.
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine.
* Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice.
* Use of an oral care product indicated for the relief of dentine hypersensitivity within 8 weeks of screening.
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain.

Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering and anti-inflammatory drugs.

* Currently taking antibiotics or has taken antibiotics within 2 weeks of Baseline.
* Daily dose of a medication which, in the opinion of the Investigator, is causing xerostomia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-03-11 (Actual); Study Completion 2016-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mississauga, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single center in Canada.
Pre-assignment Details: A total of 143 participants were enrolled in the study. Out of which 141 participants were randomized.
Groups:
- Stannous Fluoride Dentifrice: Participants were instructed to dose a dry toothbrush with a full strip of toothpaste containing 0.454% weight by weight (w/w) stannous fluoride (1100 parts per million [ppm] fluoride), then brush each of the two selected sensitive test teeth first, followed by the whole mouth thoroughly for at least 1 minute twice daily (morning and evening). Participants were permitted to rinse with tap water.
- Sodium Monofluorophosphate Dentifrice: Participants were instructed to apply a full brush head of toothpaste to a dry toothbrush containing 0.76% sodium monofluorophosphate (1000ppm fluoride), and then brush the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water.
Period: Overall Study
Arm/Group | Stannous Fluoride Dentifrice | Sodium Monofluorophosphate Dentifrice
Started | 71 | 70
Completed | 71 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant was randomized to sodium monofluorophosphate dentifrice but received stannous fluoride dentifrice, therefore, treatment arm "stannous fluoride dentifrice" included 72 participants & treatment arm "sodium monofluorophosphate dentifrice" included 69 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stannous Fluoride Dentifrice | Sodium Monofluorophosphate Dentifrice | Total
Number analyzed (Participants) | 72 | 69 | 141
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (10.27) | 48.0 (10.58) | 47.9 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 50 | 105
  Male | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score at Day 14
Description: Schiff Sensitivity Score is an examiner based index, was scored immediately following administration of the evaporative air stimulus by directing a maximum one second application of air from a dental air syringe to the exposed dentine surface from a distance of approximately 1 cm. The examiner indicated the participant's response to the evaporative air stimulus, after the stimulation of each individual tooth, using the Schiff sensitivity scale as follows: 0= participant does not respond to air stimulation; 1= participant responds to air stimulus but does not request discontinuation of stimulus; 2= participant responds to air stimulus and requests discontinuation or moves from stimulus; 3= participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Time Frame: Baseline, Day 14
Population: Analysis for this outcome was conducted on Intent-to-treat (ITT) population which included all participants who were randomized, received at least one dose of the study treatment and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stannous Fluoride Dentifrice: Participants were instructed to dose a dry toothbrush with a full strip of toothpaste, then brush each of the two selected sensitive test teeth first, followed by the whole mouth thoroughly for at least 1 minute twice daily (morning and evening). Participants were permitted to rinse with tap water.
- Sodium Monofluorophosphate Dentifrice: Participants were instructed to apply a full brush head of toothpaste to a dry toothbrush, and then brush the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water.
Arm/Group | Stannous Fluoride Dentifrice | Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 71 | 70
score on a scale
  At Baseline | 2.70 (0.427) | 2.74 (0.423)
  Change From Baseline at Day 14 | -1.38 (0.843) | -0.10 (0.405)
Statistical Analysis 1: Comparison: Stannous Fluoride Dentifrice vs Sodium Monofluorophosphate Dentifrice; Test type: Superiority or Other; p < 0.0001, ANCOVA; From ANCOVA model with change from baseline in Schiff Sensitivity Score as response and treatment and baseline Schiff sensitivity score as covariates; Least square (LS) mean difference = -1.29, 95% CI 2-sided [-1.509 to -1.071] — Difference is first named dentifrice minus second named dentifrice such that a negative difference favours first named dentifrice

2. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score at Day 7
Description: as for outcome 1
Time Frame: Baseline, Day 7
Population: Analysis for this outcome was conducted on ITT population which included all participants who were randomized, received at least one dose of the study treatment and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stannous Fluoride Dentifrice | Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 71 | 70
score on a scale
  At Baseline | 2.70 (0.427) | 2.74 (0.423)
  Change from baseline at Week 7 | -0.74 (0.446) | -0.04 (0.374)

3. Secondary Outcome: Change From Baseline in Tactile Threshold at Day 7 and Day 14
Description: A tactile stimulus was administered using a constant pressure probe (Yeaple Probe). Response to this stimulus was evaluated as tactile threshold. The constant pressure probe allowed the examiner to vary the force applied to the dentine surface from 10 g to an upper threshold of 80 g in increments of 10 g. The tactile threshold is the maximum pressure applied without the participant's reporting pain or discomfort. The greater the tactile threshold, the less sensitive the tooth.
Time Frame: Baseline, Day 7 and Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram (g)
Arm/Group | Stannous Fluoride Dentifrice | Sodium Monofluorophosphate Dentifrice
Number analyzed (Participants) | 71 | 70
gram (g)
  At Baseline | 11.83 (3.189) | 11.50 (2.992)
  Change from Baseline at Day 7 | 5.92 (6.113) | 0.86 (3.898)
  Change from Baseline at Day 14 | 15.21 (11.663) | 0.86 (3.708)

ADVERSE EVENTS:
Time Frame: From start of screening to 5 days following last administration of the study product (up to 39 days)
Description: Safety population included 72 participants in treatment arm "stannous fluoride dentifrice" & 69 participants in treatment arm "sodium monofluorophosphate dentifrice".
Groups:
- Stannous Fluoride Dentifrice: Participants were instructed to topically dose a dry toothbrush with a full strip of toothpaste, then brush each of the two selected sensitive test teeth first, followed by the whole mouth thoroughly for at least 1 minute twice daily (morning and evening). Participants were permitted to rinse with tap water.
- Sodium Monofluorophosphate Dentifrice: Participants were instructed to topically apply a full brush head of toothpaste to a dry toothbrush, then brush the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water.
Arm/Group | Stannous Fluoride Dentifrice | Sodium Monofluorophosphate Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/69
Other Adverse Events (participants affected / at risk) | 3/72 | 0/69
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stannous Fluoride Dentifrice (N=72) | Sodium Monofluorophosphate Dentifrice (N=69)
Pyrexia (General disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.